CLINICAL TRIAL: NCT06816914
Title: Perioperative NALIRIFOX (liposomal Irinotecan in Combination with Fluorouracil, Leucovorin, and Oxaliplatin) in Resectable Pancreatic Adenocarcinoma: Randomized Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other); China Medical University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsin-Chen Lin, Medical Doctor, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF24596A
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Resectable Pancreatic Adenocarcinoma
Keywords: Perioperative; NALIRIFOX; resectable pancreatic adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront surgery (Active Comparator): Patient in upfront surgery arm will receive operation followed by adjuvant chemotherapy with NALIRIFOX
  Interventions: Drug: NALIRIFOX
- Perioperative NALIRIFOX (Experimental): Patient in experimental arm will receive neoadjuvant NALIRIFOX followed by operation than adjuvant NALIRIFOX after operation.
  Interventions: Drug: NALIRIFOX

INTERVENTIONS:
Drug: NALIRIFOX — Patient in upfront surgery arm will receive operation followed by adjuvant chemotherapy with NALIRIFOX; patient in experimental arm will receive neoadjuvant NALIRIFOX followed by operation than adjuvant NALIRIFOX after operation.

SUMMARY:
To explore the safety and activity of NALIRIFOX (liposomal irinotecan in combination with fluorouracil, leucovorin, and oxaliplatin) in the perioperative and adjuvant treatment in resectable pancreatic adeneocarcinoma.

DETAILED DESCRIPTION:
Adjuvant chemotherapy after surgery significantly improved the survival of pancreatic cancer patients, but there is a problem that only about 50% of patients start adjuvant chemotherapy after pancreatectomy. Neoadjuvant chemotherapy might control potential metastatic lesion which are not being detected in early disease status and improve the R0 resection rate. Additionally, it prevents unnecessary surgeries by selecting patients with rapid disease progression. Furthermore, compared with chemotherapy administered after surgery, more patients can complete the planned chemotherapy schedule in neoadjuvant setting. NALIRIFOX was approved its efficacy and safety in metastatic pancreatic cancer, but its role in perioperative setting is unknown. In this study, we want to o explore the safety and activity of NALIRIFOX in the perioperative and adjuvant treatment in resectable pancreatic adeneocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* previously untreated, histologically or cytologically proven PDAC
* age between 20 and 75 years at registration
* ECOG performance status of 0 or 1
* AJCC (8th edition) clinical stage I or II with measurable disease (CT or MRI) in the pancreas. (positron emission tomography scan alone not allowed)
* Surgically resectable disease according to NCCN criteria (Version 1.2023 - May 4, 2023):
* no arterial tumor contact (celiac axis, superior mesentery artery, or common hepatic artery).
* no tumor contact with the superior mesentery vein or portal vein or ≤180° contact without vein contour irregularity.
* adequate major organ functions
* Women of childbearing potential (including women with chemical menopause or no menstruation for other medical reasons) must agree to use contraception from the time ofinformed consent until 6 months or more after the last dose of investigational products. Also, women must agree not to breastfeed from the time of informed consent until 6 months or more after the last dose of the investigational product.
* Men must agree to use contraception from the start of study treatment until 3 months or more after the last dose of the investigational product.
* Participants must have signed written informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

* presence of clinically significant co-morbid medical conditions within 4 weeks prior registration judged by Investigators
* severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) in past 6 months
* New York Heart Association class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure or known abnormal electrocardiogram (ECG) with clinically significant abnormal findings in past 6 months
* interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity within 28 days prior to registration
* presence of diarrhea ≥ CTCAE v.5.0 grade 2
* concomitant systemic infection requiring treatment
* prior organ allograft or allogeneic bone marrow transplantation
* known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome
* prior or concurrent malignancies within the last 3 years, with the exception of carcinoma in situ of the cervix, or basal type skin cancer
* any major surgery within 4 weeks of study treatment. Participants must have recovered from the effects of major surgery or significant traumatic injury at least 4 weeks before study treatment.
* pregnant women or nursing mothers, or positive pregnancy tests
* severe mental disorder
* current use or any use in past 2 weeks of strong cytochrome P450 3A4 enzyme inducers/inhibitors and/or strong UGT1A inhibitors
* known hypersensitivity to any of the components of study drugs

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-05 (Estimated); Primary Completion 2027-02-05 (Estimated); Study Completion 2028-02-05 (Estimated)

PRIMARY OUTCOMES:
12-month EFS rate | From enrollment to the event in 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan-Shen Shan, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (9):
- Taiwan (9):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No